CLINICAL TRIAL: NCT05345496
Title: Assessment of Central and Peripheral Sensitization, and Pain Mediators and Health Status in the Work-related Thumb Pain Among Physiotherapists. A Case-control Study Comparing Workers and Students
Brief Title: Central and Peripheral Sensitization, Pain Mediators in Thumb Pain Among Physiotherapists
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giacomo Carta, PhD Candidate Experimental Medicine and Therapy, MSc in Rehabilitation Scence, BSc in Pysiotherapy, University of Turin, Italy
Other Study IDs: 0169961-14/03/22
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Work-related Illness
Keywords: Thumb pain; Central sensistization; Peripheral sensitization; Modulating factors; ICF; Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WORKERS GROUP: 44 physiotherapists with a history of at least 1 painful episode of work-related thumb pain in the last 3 months will be enrolled.
- STUDENT GROUP: 44 physiotherapy students in their first academic year will be enrolled.

SUMMARY:
The work-related thumb pain is a common problem among physiotherapists which deal with this experience at least once in their life. Several studies analyzed the distribution of mechanical forces, kinematics, and kinesiology of the thumb in this clinical condition. However, there is no data, available in the literature, on how this pain processed is sustained and if plastic changes in the central or peripheral nervous system are involved. The research aims are to investigate the relationship between the thumb pain and pain related central and peripheral nervous sensitization phenomena among physiotherapists (exposed to work) and physiotherapy students (not exposed). The relevance of each of the pain chronification mediators, reported in the literature (anxiety, depression catastrophization, self-efficacy, kinesiophobia) will be also defined. Data on pain intensity, muscle strength, and endurance in the hand will be collected and the relation between peripheral sensitization phenomena in the hand, and central sensitization will be assessed. Also, the relevance of pain mediators and the health perceived status will be assess adopting validated questionnaires and the minimal Generic ICF core set.

DETAILED DESCRIPTION:
Introduction: Physiotherapists' work-related thumb pain is a problem recognized by the World Health Organization to be the major work-related musculoskeletal problems (WMSDs) for this profession. About 70.8% of physiotherapists experience thumb pain at least once in their life. In those who practice manual therapy, thumb pain can determine the use of compensatory strategies or the impossibility to practice wanted manipulation. It has been estimated that 1 in 6 physiotherapists end their careers because of WMSDs. The data available in the literature on biomechanics for this phenomenon do not allow to define a proper causa relation lacking to describe the impact of pain mechanisms involved, the impact of mediators of chronicity in pain, and health status.

The purpose of the present research is to investigate the relation between thumb pain and phenomena of central or peripheral plasticity among physiotherapists (exposed) and compare this data to physiotherapy students (not exposed). In particular, we aim to identify the relevance of each chronic pain mediator described in the literature (anxiety, depression, self-efficacy, kinesiophobia) in this health condition.

Methods: A case-control study will be performed. 44 physiotherapists with thumb pain and 44 physiotherapy students will be evaluated. Muscle strength and endurance of the hand will be assessed. Assessment of peripheral sensitization phenomena will be performed with validated clinical tests. It will also be assessed the health status through the minimal ICF core set, the intensity of pain, and through validated questionnaires the central sensitization, anxiety, depression, catastrophization, kinesiophobia, and self-efficacy. The sample size of 44 subjects per group (10% dropout) was estimated a priori, with a clinically relevant effect size of d= .80 and with an estimated power (1- beta )= .95 and α= 0.05.

Expected results: The results of this study can improve the knowledge of the pain mechanisms involved and the complexity of this work-related disabling condition following a multifactorial biopsychosocial model. Results could also improve the prevention of thumb pain in physiotherapists with a relevant impact on this work-related disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects giving their written consent to be enrolled in the study.
* Subjects aged more than 18 years old.
* Registration to the professional register or to the degree course in Physiotherapy
* History of at least 1 episode of work-related thumb pain in the last 3 months for physiotherapists

Exclusion Criteria:

* Recent or current pain/pathology of the upper limbs and neck;
* Pregnancy;
* Neurological disorders that increase or decrease the tone of upper limb and neck muscles;
* Rheumatic diseases
* Recent hand surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapists registered in the professional register University students in physiotherapy BSc.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Italian Central Sensitization Inventory (CSI-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be adopted to assess central sensitization. It consists of two sections. Part A is made up of 25 self-reported items, each rated on a scale from 0 to 5 (0=never and 4=always), for a maximum score of 100. Part B analyses the presence of commonly related symptoms. A total score < 40 shows good sensitivity to exclude the presence of signs and symptoms related to central sensitization.
Quantitative sensory testing (QST) | Tests will be administered on day 1 for each site, by a physiotherapist using Neuropen
  These tests will be adopted to assess peripheral and central sensitiazion phenomena.It will be tested 1cm2 of both dorsal and palmar skin. First, using the Neuropen tool patient will be asked to discriminate between a set of 3 alterante tactile and puncture stimuli. Then a mechanical pressure will be maintained on both sides for 10 seconds and asked if it was painful or not. Then 10 puncture stimuli in a row with Neuropen will be performed recording pain intensity.

SECONDARY OUTCOMES:
International Classification of Functioning, Disability, and Health Generic Core Set | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess the subject's health status. It consists in 7 items and includes the following subcategories: body functions (physiological functions of the body system), body structures (anatomical components such as organs, limbs, and their components), activities (execution of a task or activity by an individual), and participation (involvement in daily life).
Italian Pain Catastrophizing Scale (PCS-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess the catastrophization. This scale consists of 13 items divided into three domains. Each item can achieve a maximum of 4 points, for a maximum of 52. The higher the score, the greater the presence of thoughts of catastrophization.
Italian Tampa Scale for Kinesophobia (TSK-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to measure kinesiophobia and fear of movement. This scale consists of 17 items assessing the fear of movement perception, scored 1 to 4 points (1=totally disagreeing: 4= strongly agree), achieving a score that varies between 17 and 68. The higher the score, the higher the level of fear related to movement.
Italian Hospital Anxiety Depression Scale (HADS-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess anxiety and depression.This scale consists of 14 items divided into two subcategories. The first 7 items investigate General anxiety, while the other 7 items, mainly investigate the state of anhedonia. For each item the score varies from 0-3 (0= absence; 3= extreme presence). Higher scores correspond to high levels of anxiety and depression.
Italian Pain Self-efficacy Questionnaire (PSEQ-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to detect self-efficacy. This scale consists of 10 items, whose score varies from 0-6 (0=not safe at all, 10= completely safe), for a total of 60 points. The lower the score, the lower the self-efficacy is.
Upper Limb Neural Tension Test (ULNTT 1) | the test will be administered on day 1 by a physiotherapist during the clinical examination
  It will be used to assess mechanosensitivity of the brachial plexus and upper limb nerves. It consists of a validated combination of physiological movement of the arm (shoulder depression, wrist and finger extension, forearm supination, shoulder external rotation, and elbow extension) and a symptom discrimination maneuvers (homolateral and contralateral cervical spine inclination) to assess the physiological mechanosensitivity of the nerves of the upper limb.
Vagus nerve neurodynamic test (VN-NDT) | the test will be administered on day 1 by a physiotherapist during the clinical examination
  It will be performed to assess vagus nerve sensitization due to chronic stress. It consists of a combination of physiological movements of the neck (upper cervical flexion, contralateral lateral flexion, ipsilateral rotation) and gentle movements of the upper abdomen caudally and cranially to increase tension on the thoracic tract of the vagus nerve, and it assess the physiological mechanosensitivity of the vagus nerve and its effects on heart rate at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, MSc, PT BSc, Principal Investigator — University of Turin, Italy
Locations (1):
- Department of Biological and Clinical Science - University of Turin, Orbassano, TO, Italy

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All of the individual particiapnt data collected during the trial will be shared after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following the publication. No end date.
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.